CLINICAL TRIAL: NCT00633490
Title: Phase 1 Study of Apatinib as an Inhibitor of Angiogenesis
Brief Title: Study of Apatinib as an Inhibitor of Tumor Angiogenesis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Jin Li/Dr, Fudan University cancer hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007APA
Record Dates: First submitted 2008-02-24; First posted 2008-03-12 (Estimated); Last update posted 2008-07-22 (Estimated); Status verified 2008-03

CONDITIONS: Tumor
Keywords: Toxicity; Efficacy
MeSH Terms: conditions — Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: apatinib

INTERVENTIONS:
Drug: apatinib — apatinib is a tablet in the form of 250mg and 100mg and 50mg, orally, daily
  Other Names: mesylate apatinib

SUMMARY:
Apatinib is a tyrosin-inhibitor agent targeting at vascular endothelial growth factor receptor (VEGFR), so it can inhibit tumor angiogenesis. This phase I study aims to determine the drug's toxicity and to find a dose level to be used in a phase II study in solid tumor patients.

DETAILED DESCRIPTION:
Apatinib is a tyrosin-inhibitor agent targeting at VEGFR (vasoendothelial growth factor receptor) to inhibit tumor angiogenesis. The anti-angiogenesis effect of apatinib has been viewed in preclinical tests (see protocol). This phase I clinical study is going to evaluate its toxicity and to find an appropriate dose level to be used in a phase II study in heavily treated solid tumor patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 70 years of age
* Histological or cytological confirmed solid malignant tumor
* ECOG performance status of ≤ 2
* Standard regimen failed or no standard regimen available
* Life expectancy of more than 3 months
* Duration from the last therapy is more than 6 weeks for nitroso or mitomycin; more than 4 weeks for operation or radiotherapy; more than 4 weeks for cytotoxic agents or growth inhibitors.
* Laboratory values: hemoglobin ≥ 9.0g/dl, neutrophils ≥ 1.5×10^9/L, platelets ≥ 100×10^9/L , ALT ≤ 2.5 x upper limit of normal (ULN), AST ≤ 2.5 x ULN, serum bilirubin ≤ 1.5 x ULN, serum creatine ≤ 1.5 x ULN, creatinine clearance rate ≥ 50ml/min, PT, APTT, TT, Fbg normal

Exclusion Criteria:

* Pregnant or lactating women
* Any factors that influence the usage of oral administration
* Evidence of CNS metastasis
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Intercurrence with one of the following: hypertension, coronary artery disease, arrhythmia and heart failure
* Receiving the therapy of thrombolysis or anticoagulation
* Abuse of alcohol or drugs
* Allergy to the ingredient of the agent or more than two kinds of food and drug
* Less than 4 weeks from the last clinical trial
* Disability of serious uncontrolled intercurrence infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
toxicity and tolerable dosage on the basis of NCI-CTCAE 3.0 | 4 weeks

SECONDARY OUTCOMES:
efficacy | every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li J, Zhao X, Chen L, Guo H, Lv F, Jia K, Yv K, Wang F, Li C, Qian J, Zheng C, Zuo Y. Safety and pharmacokinetics of novel selective vascular endothelial growth factor receptor-2 inhibitor YN968D1 in patients with advanced malignancies. BMC Cancer. 2010 Oct 5;10:529. doi: 10.1186/1471-2407-10-529. PMID 20923544